CLINICAL TRIAL: NCT00002679
Title: Sequential Adjuvant Chemotherapy With Doxorubicin, Taxol, and Cyclophosphamide for Stage II or III Resectable Breast Cancer With Four or More Involved Axillary Lymph Nodes
Brief Title: Adjuvant High-Dose, Sequential Chemotherapy in Treating Patients With Resected Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Maysa Abu-Khalaf, MD, Principal Investigator, Yale University School of Medicine
Purpose: Treatment
Other Study IDs: CDR0000064337; YALE-HIC-7374; NCI-V95-0720
Record Dates: First submitted 1999-11-01; First posted 2004-02-06 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Filgrastim; Cyclophosphamide; Doxorubicin; Paclitaxel; Tamoxifen; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Drug: tamoxifen citrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose sequential chemotherapy as adjuvant therapy in treating patients with stage II or stage III breast cancer who have four or more positive axillary lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of dose intensive, sequential adjuvant chemotherapy with doxorubicin, paclitaxel, and cyclophosphamide in patients with stage II/III resected breast cancer. II. Evaluate the toxicity of this regimen in these patients.

OUTLINE: All patients receive sequential chemotherapy regimens consisting of 3 courses each of doxorubicin, paclitaxel, and cyclophosphamide on a schedule of one course every 14 days. Following completion of chemotherapy, patients who underwent breast conservation surgery receive radiotherapy. Mastectomy patients with 10 or more positive nodes or with T3-4 tumors are also eligible for delayed radiotherapy. Patients who are hormone receptor positive (or whose receptor status is unknown) are treated with oral tamoxifen for 5 years, beginning after completion of all other therapy. Patients are followed every 3 months for 2 years, every 6 months for 3 years, then yearly.

PROJECTED ACCRUAL: At total of 90 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the breast with involvement of 4 or more axillary nodes, including any T N1 M0 Concurrent bilateral breast cancer allowed Complete resection required Total mastectomy or breast conserving surgery Adjuvant radiotherapy planned after protocol chemotherapy Clear surgical margins Axillary dissection yielding at least 9 lymph nodes Entry required within 8 weeks of definitive surgery Hormone receptor status: Any status

PATIENT CHARACTERISTICS: Age: Over 18 Sex: Not specified Menopausal status: Not specified Performance status: Karnofsky 80%-100% ECOG 0 or 1 Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 times normal AST no greater than 2 times normal Alkaline phosphatase no greater than 2 times normal Renal: Creatinine no greater than 1.8 mg/dL OR Creatinine clearance at least 60 mL/min Urinalysis normal Cardiovascular: Left ventricular ejection fraction normal on MUGA or echocardiogram No congestive heart failure requiring medical therapy No serious arrhythmia No first-, second-, or third-degree heart block Other: No abnormal CT of chest or abdomen No uncontrolled infection No serious medical condition that would prevent treatment No second malignancy except curatively treated: Nonmelanomatous skin cancer Carcinoma in situ of the cervix Not pregnant Negative pregnancy test Barrier contraception required of fertile patients before, during, and for 6 months after protocol therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior systemic chemotherapy Endocrine Therapy: No concurrent hormonal therapy unless unrelated to cancer Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: No concurrent medication affecting conduction unless cleared by a cardiologist, e.g.: Beta blockers Digoxin Antiarrhythmia agents Calcium channel blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 1994-02; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khalaf, MD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States